CLINICAL TRIAL: NCT06627413
Title: A Phase 1b, Open-label Study to Determine the Pharmacokinetics, Safety, and Tolerability of Single, Ascending Doses of Lumateperone Long-acting Injectable Formulations Administered Intramuscularly to Patients With Schizophrenia or Schizoaffective Disorder
Brief Title: Safety, Tolerability, and Pharmacokinetics of Lumateperone Long-Acting Injectable Formulations in Patients With Schizophrenia or Schizoaffective Disorder
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Intra-Cellular Therapies, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ITI-007-037
Record Dates: First submitted 2024-10-02; First posted 2024-10-04 (Actual); Last update posted 2025-03-24 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia or Schizoaffective
MeSH Terms: conditions — Schizophrenia | interventions — lumateperone

STUDY DESIGN:
Intervention Model Description: This study includes 3 sequential study parts (Parts A, B and C). Part A consists of 4 cohorts (Cohorts 1 to 4), Part B of up to 3 cohorts (Cohorts 5 to 7), and Part C of up to 2 cohorts (Cohorts 8 and 9). Within each study part, cohorts may be enrolled in parallel.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (9):
- Cohort 1 (Experimental): Lumateperone 42 mg once daily for 5 days following by a single IM dose of lumateperone 100 mg LAI formulation X500-E2 after a 5-day washout
  Interventions: Drug: Lumateperone Capsule; Drug: Lumateperone LAI
- Cohort 2 (Experimental): Lumateperone 42 mg once daily for 5 days following by a single IM dose of lumateperone 100 mg LAI formulation X500-E3 after a 5-day washout
  Interventions: Drug: Lumateperone Capsule; Drug: Lumateperone LAI
- Cohort 3 (Experimental): Lumateperone 42 mg once daily for 5 days following by a single IM dose of lumateperone 100 mg LAI formulation X500-X2 after a 5-day washout
  Interventions: Drug: Lumateperone Capsule; Drug: Lumateperone LAI
- Cohort 4 (Experimental): Lumateperone 42 mg once daily for 5 days following by a single IM dose of lumateperone 100 mg LAI formulation X500-X5 after a 5-day washout
  Interventions: Drug: Lumateperone Capsule; Drug: Lumateperone LAI
- Cohort 5 (Experimental): Lumateperone 42 mg once daily for 5 days following by a single IM dose (> 100 mg) of lumateperone LAI formulation (chosen from Part A) after a 5-day washout
  Interventions: Drug: Lumateperone Capsule; Drug: Lumateperone LAI
- Cohort 6 (Experimental): Lumateperone 42 mg once daily for 5 days following by a single IM dose (> 100 mg) of lumateperone LAI formulation (chosen from Part A) after a 5-day washout
  Interventions: Drug: Lumateperone Capsule; Drug: Lumateperone LAI
- Cohort 7 (Experimental): Lumateperone 42 mg once daily for 5 days following by a single IM dose (> 100 mg) of lumateperone LAI formulation (chosen from Part A) after a 5-day washout
  Interventions: Drug: Lumateperone Capsule; Drug: Lumateperone LAI
- Cohort 8 (Experimental): Lumateperone 42 mg once daily for 5 days following by a single IM dose (> dose in Part B) of lumateperone LAI formulation (chosen from Part B) after a 5-day washout
  Interventions: Drug: Lumateperone Capsule; Drug: Lumateperone LAI
- Cohort 9 (Experimental): Lumateperone 42 mg once daily for 5 days following by a single IM dose (> dose in Part B) of lumateperone LAI formulation (chosen from Part B) after a 5-day washout
  Interventions: Drug: Lumateperone Capsule; Drug: Lumateperone LAI

INTERVENTIONS:
Drug: Lumateperone Capsule — Lumateperone 42 mg capsule, oral administration
Drug: Lumateperone LAI — Lumateperone LAI X500-E2 IM injection
  Arms: Cohort 1
Drug: Lumateperone LAI — Lumateperone LAI X500-E3 IM injection
  Arms: Cohort 2
Drug: Lumateperone LAI — Lumateperone LAI X500-X2 IM injection
  Arms: Cohort 3
Drug: Lumateperone LAI — Lumateperone LAI X500-X5 IM injection
  Arms: Cohort 4
Drug: Lumateperone LAI — Lumateperone LAI (X500-E2 or X500-E3 or X500-X2 or X500-X5) IM injection
  Arms: Cohort 5; Cohort 6; Cohort 7; Cohort 8; Cohort 9

SUMMARY:
Study ITI-007-037 is a Phase 1b, open-label study to evaluate the safety, tolerability, and PK of lumateperone long-acting injectable (LAI) formulations after a single intramuscular injection in patients with stale schizophrenia or schizoaffective disorder.

ELIGIBILITY:
Main Inclusion Criteria:

* Male or female patients between 18 and 55 years of age, inclusive;
* Clinical diagnosis of schizophrenia or schizoaffective disorder according to Diagnostic and Statistical Manual of Mental Disorders (DSM-5);
* Clinically stable and free from acute exacerbation of psychosis for at least 3 months prior to Screening;
* Clinical Global Impression - Severity (CGI-S) score ≤ 3 at Screening and prior to dosing on Day 1;
* Body mass index (BMI) between 18.0 and 38.0 kg/m2, inclusive at Screening, and a minimum body weight of 50 kg at Screening.

Main Exclusion Criteria:

* History of psychiatric condition other than schizophrenia that, in the Investigator's opinion, may be detrimental to participation in the study;
* Any suicidal ideation or wish to be dead within the past 6 months of Screening, any suicide attempt within the past 2 years prior to Screening, or any current concern for the patient's safety based on the Columbia-Suicide Severity Rating Scale (C-SSRS) (excluding self-injurious, non-suicidal behavior), and/or Investigator assessment that the patient is a safety risk to him/herself or others;
* Clinically significant abnormality within 2 years of Screening that in the Investigator's opinion may place the patient at risk or interfere with study outcome variables;
* Has a QT interval corrected for heart rate using Fridericia formula > 450 msec in males or > 470 msec in females, or evidence of clinically significant bundle branch blocks on ECG at Screening.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 72 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Pharmacokinetics: Cmax,oral | Day 5
  Maximum plasma concentration of lumateperone
Pharmacokinetics: Cmax,IM | Day 11-60
  Maximum plasma concentration of lumateperone
Pharmacokinetics: Tmax,oral | Day 5
  Time of maximum concentration of lumateperone in plasma
Pharmacokinetics: Tmax,IM | Day 11-60
  Time of maximum concentration of lumateperone in plasma
Pharmacokinetics: AUC0-t,oral | Day 5
  Area under the plasma concentration time curve from time zero to the last measurable of concentration of lumateperone
Pharmacokinetics: AUC0-t,IM | Day 11-60
  Area under the plasma concentration time curve from time zero to the last measurable of concentration of lumateperone

SECONDARY OUTCOMES:
Percentage of subjects with treatment-emergent adverse events | up to 30 days after the last protocol-defined study visit
Change from baseline in systolic and diastolic blood pressure | Days 25 and 60
Change from baseline in ECG QTcF interval | Days 25 and 60
Change from baseline in hemoglobin | Days 25 and 60
Change from baseline in white blood cell count | Days 25 and 60
Change from baseline in aspartate aminotransferase | Days 25 and 60
Change from baseline in alanine aminotransferase | Days 25 and 60
Change from baseline in Abnormal Involuntary Movement Scale (AIMS) | Days 25 and 60
  AIMS is a measure of facial and oral movements, extremity movements and trunk movements. Items are rated on a scale from none (0) to severe (4).

CONTACTS AND LOCATIONS:
Locations (4):
- United States (4):
  - Clinical Site 2, Los Alamitos, California
  - Clinical Site 3, Atlanta, Georgia
  - Clinical Site 4, Decatur, Georgia
  - Clinical Site 1, Marlton, New Jersey